CLINICAL TRIAL: NCT05401812
Title: A Factorial Trial of Glucocorticoid Therapy in Acute Respiratory Distress Syndrome: Optimizing Dosing Regimen and Developing Biomarker-guided Treatment
Brief Title: Glucocorticoid Therapy for Acute Respiratory Distress Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult enrollment
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 202012189MINB
Record Dates: First submitted 2022-01-02; First posted 2022-06-02 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Corticosteroid; Glucocorticoid
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Standard care without glucocorticoid therapy.
- Low dose and long treatment duration (Experimental): Methylprednisolone equivalent dose 0.5 mg/kg/day for 5 days, followed by 0.25 mg/kg/day for 5 days.
  Interventions: Drug: Intravenous glucocorticoid therapy
- Low dose and short treatment duration (Experimental): Methylprednisolone equivalent dose 0.5 mg/kg/day for 4 days,, followed by 0.25 mg/kg/day for 3 days.
  Interventions: Drug: Intravenous glucocorticoid therapy
- Moderate dose and long treatment duration (Experimental): Methylprednisolone equivalent dose 1 mg/kg/day for 5 days, followed by 0.5 mg/kg/day for 5 days.
  Interventions: Drug: Intravenous glucocorticoid therapy
- Moderate dose and short treatment duration (Experimental): Methylprednisolone equivalent dose 1 mg/kg/day for 4 days, followed by 0.5 mg/kg/day for 3 days.
  Interventions: Drug: Intravenous glucocorticoid therapy

INTERVENTIONS:
Drug: Intravenous glucocorticoid therapy — Betamethasone, dexamethasone, or methylprednisolone
  Arms: Low dose and long treatment duration; Low dose and short treatment duration; Moderate dose and long treatment duration; Moderate dose and short treatment duration

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a clinical syndrome of inflammatory lung injury characterized by increased pulmonary vascular permeability, loss of aerated lung tissue, severe hypoxemia and impaired compliance. Despite the advance in the critical care technology, the mortality of ARDS remains high in the last decades. Glucocorticoids have profound anti-inflammatory actions through the pleiotropic effects of the glucocorticoid receptor, which are considering a promising pharmacological therapy to mitigate the inflammatory lung injury and subsequent fibrosis in ARDS. Previous clinical trials have repeatedly tested the efficacy of glucocorticoid therapy in ARDS; however, the data about hard outcomes, such as mortality, are inconsistent between these studies. Investigators designed a 3x2 factorial trial of glucocorticoid therapy in ARDS to test the effects of glucocorticoid dosages (dose 0, dose 0.5 mg/kg, and dose 1 mg/kg of methylprednisolone equivalence) and durations (prolonged and short duration) on the treatment efficacy. In addition, investigators will measure the change of inflammatory biomarkers for post-hoc analysis to explore whether biomarkers could be used to guide patient selection and steroid tapering.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe ARDS with a P/F ratio < 200 mmHg
2. On invasive mechanical ventilation
3. The onset of ARDS < 72 hours

Exclusion Criteria:

1. Age <20 years
2. Receiving systemic glucocorticoid therapy
3. Uncontrolled gastrointestinal bleeding
4. Terminal cancer
5. Post-operation or with large wound
6. Considered by the primary care doctor to be either definitely indicated or definitely contraindicated for glucocorticoid therapy
7. Anticipating to receive chemotherapy and immunotherapy in 3 months
8. Uncontrolled fungal infection
9. Post solid organ or bone marrow transplant
10. Severe influenza without anti-viral therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free survival | 28 days
  Ventilator-free survival between control and intervention arms

SECONDARY OUTCOMES:
Glucocorticoid dose and ventilator-free survival | 28 days
  Ventilator-free survival between low-dose and moderate-dose glucocorticoid groups
Glucocorticoid treatment duration and ventilator-free survival | 28 days
  Ventilator-free survival between long treatment duration and short treatment duration groups
ICU mortality | Length of ICU stay up to 28 days
  Between-group difference in mortality at ICU discharge
Hospital mortality | Length of hospital stay up to 60 days
  Between-group difference in mortality at hospital discharge
60-day mortality | 60 days
  Between-group difference in mortality by day 60
Oxygenation on day 7 | 7 days
  Proportion of patients with a P/F ratio > 200 mmHg on day 7
Rapid oxygenation improvement | 3 days
  Change in P/F ratios between day 1 and day 3
Successful liberation from mechanical ventilation | Up to 60 days
  Median time to successful liberation from mechanical ventilation
Lymphocytopenia | 7 days
  Proportion of lymphocytopenia on day 7
Blood glucose level | 10 days
  Peak blood glucose level during treatment
Hyperglycemia | 10 days
  Proportion of patients with hyperglycemia during treatment

IPD SHARING:
Plan to Share IPD: Undecided